CLINICAL TRIAL: NCT04851054
Title: Postoperative Serum VEGF Concentration as an Independent Prognostic Factor for Recurrence After Curative Colon Cancer Surgery. Multicentric Study.
Brief Title: Postoperative VEGF and Recurrence After Colon Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital del Mar (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Hospital de Granollers (Other); Althaia Xarxa Assistencial Universitària de Manresa (Other); Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Marta Pascual, CHIEF, COLON AND RECTAL SURGERY, DEPARTMEN OF SURGERY, Hospital del Mar
Other Study IDs: 2015/6097/I
Record Dates: First submitted 2021-03-11; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Angiogenesis; Colon Cancer; Surgery; Recurrence; VEGF Overexpression
Keywords: VEGF; Colon Cancer; Surgery; Recurrence
MeSH Terms: conditions — Colonic Neoplasms; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum samples stored at -80ºC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after surgery for colon cancer with intention to cure: Patients with colon cancer admitted to the Colorectal Surgery Unit of the centers participating in the study, who will undergo elective surgical resection with potentially curative intention
  Interventions: Procedure: Surgery for colon cancer with intention to cure

INTERVENTIONS:
Procedure: Surgery for colon cancer with intention to cure — Surgery by open or laparoscopic approach

SUMMARY:
The purpose of this trial is to study the relationship between the angiogenic response to surgical aggression, determined through the serum levels of vascular endothelial growth factor (VEGF) on postoperative day four, and the tumor recurrence in patients with colon cancer operated with a curative intention.

DETAILED DESCRIPTION:
DESIGN: Prospective multicentric study.

PARTICIPATION: Colorectal Surgery Units of Hospital del Mar, Barcelona; Hospital Universitari Joan XXIII, Tarragona; Hospital Universitari La Fe, Valencia; Hospital Clínico San Carlos, Madrid; Hospital General de Granollers, Granollers; Hospital Germans Trias i Pujol, Badalona; Athalaia, Xarxa Assistencial Universitària de Manresa, Manresa

STUDY SUBJECTS: 280 consecutive patients with non-metastatic colon cancer in whom a curative intent resection is performed.

DETERMINATIONS: Determination of the proangiogenic cytokine VEGF in serum on the postoperative day four to assess its relationship with oncological results on long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colon cancer admitted to the Colorectal Surgery Unit of the centers participating in the study,
* Patients who will undergo elective surgical resection with potentially curative intention

Exclusion Criteria:

* Patients with metastatic disease
* Patients with synchronous colon neoplasia or in the previous five years
* Patients undergoing emergency surgery
* Patients who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer admitted to the Colorectal Surgery Unit of the centers participating in the study, who will undergo elective surgical resection with potentially curative intention.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
VEGF in serum on postop day 4 | Postoperative day 4
  A 10cc sample of peripheral blood will be drawn on postoperative day 4

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL PERA, PhD, Study Chair — Hospital del Mar

IPD SHARING:
Plan to Share IPD: No